CLINICAL TRIAL: NCT02730299
Title: A Multicenter, Randomized, Phase III Registration Trial of Transplantation of NiCord®, Ex Vivo Expanded, UCB-derived, Stem and Progenitor Cells, vs. Unmanipulated UCB for Patients With Hematological Malignancies
Brief Title: Stem Cell Transplantation With NiCord® (Omidubicel) vs Standard UCB in Patients With Leukemia, Lymphoma, and MDS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gamida Cell ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GC P#05.01.020
Record Dates: First submitted 2016-03-28; First posted 2016-04-06 (Estimated); Results first posted 2022-10-25 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Hematological Malignancies; Acute Lymphoblastic Leukemia (ALL); Acute Myelogenous Leukemia (AML); Chronic Myelogenous Leukemia (CML); Myelodysplastic Syndrome (MDS); Lymphoma; Acute Leukemia
MeSH Terms: conditions — Hematologic Neoplasms; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- NiCord® (omidubicel) (Experimental): NiCord® is a cryopreserved stem/progenitor cell based product comprised of:
  1. ex vivo expanded, umbilical cord blood-derived hematopoietic CD34+ progenitor cells (NiCord® cultured fraction (CF))
  2. the non-cultured cell fraction of the same Cord Blood Unit (CBU) (NiCord® Non-cultured Fraction (NF)) consisting of mature myeloid and lymphoid cells.
  Both fractions, i.e. NiCord® CF and NiCord® NF, will be kept frozen until they are thawed and infused on the day of transplantation.
  Interventions: Drug: NiCord® (omidubicel)
- Unmanipulated CBU(s) (Active Comparator)
  Interventions: Other: Cord Blood Unit

INTERVENTIONS:
Drug: NiCord® (omidubicel)
  Arms: NiCord® (omidubicel)
Other: Cord Blood Unit — Cord blood unit
  Arms: Unmanipulated CBU(s)

SUMMARY:
This study is an open-label, controlled, multicenter, international, Phase III, randomized study of transplantation of NiCord® versus transplantation of one or two unmanipulated, unrelated cord blood units in patients with acute lymphoblastic leukemia or acute myeloid leukemia, myelodysplastic syndrome, chronic myeloid leukemia or lymphoma, all with required disease features rendering them eligible for allogeneic transplantation.

DETAILED DESCRIPTION:
Successful blood and marrow transplantation (BMT) requires the infusion of a sufficient number of hematopoietic stem/progenitor cells (HSPCs), capable of both homing to the bone marrow and regenerating a full array of hematopoietic cell lineages with early and late repopulating ability in a timely fashion.

A major drawback of Umbilical Cord Blood (UCB) is the low stem cell dose available for transplantation, compared to mobilized peripheral blood (PB) or bone marrow. This low stem cell dose can compromise the chances of engraftment and contributes to delayed kinetics of neutrophil and platelet recovery, as well as other transplant outcomes.

The aim of ex vivo expansion of cord blood is to provide a graft with sufficient numbers of cells that have rapid and robust in vivo neutrophil and platelet producing potential to enable successful transplantation.

NiCord® is a stem/progenitor cell-based product composed of ex vivo expanded allogeneic cells from one entire unit of UCB. NiCord® utilizes the small molecule nicotinamide (NAM), as an epigenetic approach to inhibit differentiation and to increase the migration, bone marrow (BM) homing and engraftment efficiency of Hematopoietic Progenitor Cells (HPC) expanded in ex vivo cultures. The chief aim of the study is to compare the safety and efficacy of NiCord® single ex-vivo expanded cord blood unit transplantation to unmanipulated cord blood unit transplantation in patients with hematological malignancies following conditioning therapy.

ELIGIBILITY:
Inclusion Criteria:

* Applicable disease criteria
* Patients must have one or two partially HLA-matched CBUs
* Back-up stem cell source
* Adequate Karnofsky/Lansky Performance score
* Sufficient physiological reserves
* Signed written informed consent

Exclusion Criteria:

* HLA-matched donor able to donate
* Prior allogeneic HSCT
* Other active malignancy
* Active or uncontrolled infection
* Active/symptoms of central nervous system (CNS) disease
* Pregnancy or lactation

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2025-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Horwitz, MD, Study Chair — Duke University
Locations (52):
- United States (21):
  - UCLA, Los Angeles, California
  - City of Hope, Los Angeles, California
  - Stanford University Cancer Institute, Palo Alto, California
  - UC San Diego Moores Cancer Center, San Diego, California
  - Children's Hospital Colorado, Denver, Colorado
  - Northwestern University, Evanston, Illinois
  - Loyola University, Cardinal Bernardin Cancer Center, Maywood, Illinois
  - University of Kansas Cancer Center, Westwood, Kansas
  - The University of Maryland Medicine Center, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Medical Center, Detroit, Michigan
  - University of Minnesota Masonic Cancer Center, Minneapolis, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic Children's, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - UPMC Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - West Cancer Clinic, Germantown, Tennessee
  - Children's Medical Center of Dallas, Dallas, Texas
  - University of Virginia Cancer Center, Charlottesville, Virginia
- Brazil (5):
  - Instituto Nacional de Câncer José Alencar Gomes da Silva - INCA, Rio de Janeiro
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo Pediatrics, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo, São Paulo
  - Hospital das Clínicas da Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
- Robert Debré, Paris, France
- Israel (6):
  - Rambam, Haifa
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - Dana-Dwek Children's Hospital, Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Chaim Sheba Medical Center, The Edmond and Lily Safra Children's hospital, Tel Litwinsky
- Italy (2):
  - Careggi University Hospital, Florence
  - Ospedale Pediatrico Bambino Gesù, Rome
- Netherlands (2):
  - University Medical Center Utrecht, Utrecht
  - Prinses Maxima Centrum voor Kinderoncologie B.V., Utrecht
- Instituto Português de Oncologia de Lisboa Francisco Gentil, Lisbon, Portugal
- Singapore (2):
  - National University Cancer Institute, Singapore
  - Singapore General Hospital, Singapore
- Spain (8):
  - Hospital Universitari Vall d'Hebron pediatrics, Barcelona
  - University Hospital Vall d'Hebron, Barcelona
  - ICO Bellvitge, Barcelona
  - Sant Joan de Deu, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Virgen del Rocío, Seville
  - Hospital Universitario La Fe, Valencia
  - Hospital Universitario y Politécnico La Fe (pediatric), Valencia
- United Kingdom (4):
  - The Royal Marsden NHS Foundation Trust, Sutton, Surrey
  - Queen Elizabeth Hospital, Birmingham
  - St James Hospital, Leeds
  - Manchester University NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Majhail NS, Miller B, Dean R, Manghani R, Shin H, Sivaraman S, Maziarz RT. Hospitalization and Healthcare Resource Utilization of Omidubicel-Onlv versus Umbilical Cord Blood Transplantation for Hematologic Malignancies: Secondary Analysis from a Pivotal Phase 3 Clinical Trial. Transplant Cell Ther. 2023 Dec;29(12):749.e1-749.e5. doi: 10.1016/j.jtct.2023.09.004. Epub 2023 Sep 12. PMID 37703995
- [Derived] Szabolcs P, Mazor RD, Yackoubov D, Levy S, Stiff P, Rezvani A, Hanna R, Wagner J, Keating A, Lindemans CA, Karras N, McGuirk J, Hamerschlak N, Lopez-Torija I, Sanz G, Valcarcel D, Horwitz ME. Immune Reconstitution Profiling Suggests Antiviral Protection after Transplantation with Omidubicel: A Phase 3 Substudy. Transplant Cell Ther. 2023 Aug;29(8):517.e1-517.e12. doi: 10.1016/j.jtct.2023.04.018. Epub 2023 Apr 28. PMID 37120136
- [Derived] Horwitz ME, Stiff PJ, Cutler C, Brunstein C, Hanna R, Maziarz RT, Rezvani AR, Karris NA, McGuirk J, Valcarcel D, Schiller GJ, Lindemans CA, Hwang WYK, Koh LP, Keating A, Khaled Y, Hamerschlak N, Frankfurt O, Peled T, Segalovich I, Blackwell B, Wease S, Freedman LS, Galamidi-Cohen E, Sanz G. Omidubicel vs standard myeloablative umbilical cord blood transplantation: results of a phase 3 randomized study. Blood. 2021 Oct 21;138(16):1429-1440. doi: 10.1182/blood.2021011719. PMID 34157093
- [Derived] Del Pozo Martin Y. 47th Annual Meeting of the EBMT. Lancet Haematol. 2021 May;8(5):e317-e318. doi: 10.1016/S2352-3026(21)00104-6. Epub 2021 Mar 31. No abstract available. PMID 33811823

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 125 patients were screened, met inclusion criteria and were randomized to treatment from 33 transplant centers worldwide. First patient was consented on 20th December 2016 and the last patient consented on 27th December 2019.
Groups:
- NiCord® (Omidubicel): NiCord® is a cryopreserved stem/progenitor cell based product comprised of:
  1. ex vivo expanded, umbilical cord blood-derived hematopoietic CD34+ progenitor cells (NiCord® cultured fraction (CF))
  2. the non-cultured cell fraction of the same Cord Blood Unit (CBU) (NiCord® Non-cultured Fraction (NF)) consisting of mature myeloid and lymphoid cells.
  Both fractions, i.e. NiCord® CF and NiCord® NF, will be kept frozen until they are thawed and infused on the day of transplantation.
  NiCord® (omidubicel)
- Unmanipulated CBU(s): Unmanipulated cord blood unit(s)
Period: Overall Study
Arm/Group | NiCord® (Omidubicel) | Unmanipulated CBU(s)
Started | 62 | 63
Completed | 62 | 63
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NiCord® (Omidubicel) | Unmanipulated CBU(s) | Total
Number analyzed (Participants) | 62 | 63 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8 | 6 | 14
  Between 18 and 65 years | 54 | 57 | 111
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 23 | 53
  Male | 32 | 40 | 72
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 6 | 16
  Not Hispanic or Latino | 46 | 52 | 98
  Unknown or Not Reported | 6 | 5 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 7 | 10 | 17
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 11 | 9 | 20
  White | 35 | 37 | 72
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 6 | 5 | 11
Region of Enrollment [Number; unit: participants]
  Netherlands | 3 | 3 | 6
  Singapore | 4 | 5 | 9
  United States | 42 | 45 | 87
  Brazil | 3 | 1 | 4
  United Kingdom | 1 | 1 | 2
  Israel | 1 | 1 | 2
  Spain | 8 | 7 | 15

OUTCOME MEASURES:

1. Primary Outcome: Time to Neutrophil Engraftment
Description: The time to engraftment of neutrophils >500/μl was defined as per Center for International Blood and Marrow Transplant Research (CIBMTR) standards, requiring donor chimerism for neutrophil engraftment.
Time Frame: post-transplant up to 42 days
Population: intent to treat
Measure: Median (95% Confidence Interval); unit: days
Groups:
- NiCord® (Omidubicel): NiCord® (omidubicel) is a cryopreserved stem/progenitor cell based product comprised of:
  1. ex vivo expanded, umbilical cord blood-derived hematopoietic CD34+ progenitor cells (cultured fraction (CF)
  2. the non-cultured cell fraction of the same Cord Blood Unit (CBU) Non-cultured Fraction (NF) consisting of mature myeloid and lymphoid cells.
- Unmanipulated Cord Blood Unit(s): Cord blood unit: Cord blood unit 1-2 units
Arm/Group | NiCord® (Omidubicel) | Unmanipulated Cord Blood Unit(s)
Number analyzed (Participants) | 62 | 63
days | 12 [10 to 14] | 22 [19 to 25]

2. Secondary Outcome: First Grade 2/3 Bacterial or Invasive Fungal Infections by 100 Days Following Transplantation
Description: First Bacterial Infection Grades 2-3 or Invasive Fungal Infection by 100 Days following Transplantation for the Intent to Treat Population
Time Frame: 100 days post-transplant
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | NiCord® (Omidubicel) | Unmanipulated CBU(s)
Number analyzed (Participants) | 62 | 63
Participants | 24 | 38

3. Secondary Outcome: Days Alive and Out of Hospital in the First 100 Days Post-transplantation
Description: Days alive and out of hospital in the first 100 Days post-transplantation for the Intent to Treat Population
Time Frame: 100 days post-transplantation
Population: Intent to Treat Population
Measure: Median (Full Range); unit: Days
Arm/Group | NiCord® (Omidubicel) | Unmanipulated CBU(s)
Number analyzed (Participants) | 62 | 63
Days | 60.5 [0 to 89] | 48 [0 to 79]

4. Secondary Outcome: Number of Participants With Platelet Engraftment by 42 Days Post-transplantation
Description: Platelet engraftment defined as the first day of a minimum of three consecutive measurements on different days such that the patient has achieved a platelet count > 20 × 10^9/L with no platelet transfusions during the preceding seven days (counting day of engraftment as one of the preceding seven days) for the Intent to Treat Population
Time Frame: 42 days post-transplantation
Population: Intent to Treat Population
Measure: Count of Participants; unit: Participants
Arm/Group | NiCord® (Omidubicel) | Unmanipulated CBU(s)
Number analyzed (Participants) | 62 | 63
Participants | 34 | 22

ADVERSE EVENTS:
Time Frame: 1 year
Description: Safety population (N=108). Serious Adverse Events (SAEs) & Adverse Events (AEs) relate to safety population (SP) (N=108).
Groups:
- Omidubicel: omidubicel is a cryopreserved stem/progenitor cell based product comprised of:
  1. ex vivo expanded, umbilical cord blood-derived hematopoietic CD34+ progenitor cells (cultured fraction (CF)
  2. the non-cultured cell fraction of the same Cord Blood Unit (CBU) Non-cultured Fraction (NF) consisting of mature myeloid and lymphoid cells.
Arm/Group | Omidubicel | Unmanipulated CBU(s)
All-Cause Mortality (participants affected / at risk) | 12/52 | 20/56
Serious Adverse Events (participants affected / at risk) | 47/52 | 51/56
Other Adverse Events (participants affected / at risk) | 52/52 | 56/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omidubicel (N=52) | Unmanipulated CBU(s) (N=56)
Febrile Neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) | 4 (4)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 2 (2)
Pyrexia (General disorders) | 5 (5) | 3 (3)
Veno-occlusive liver disease (Hepatobiliary disorders) | 2 (2) | 4 (4)
Graft-versus-host disease (Immune system disorders) | 17 (18) | 14 (15)
Femoral Neck Failure (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Transplant Failure (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
CNS events (Nervous system disorders) | 4 (4) | 2 (2)
Renal disorders (Renal and urinary disorders) | 7 (7) | 5 (5)
Respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 8 (8) | 15 (15)
GI Disorders (Gastrointestinal disorders) | 6 (6) | 13 (13)
Infections (Infections and infestations) | 26 (29) | 28 (31)
Metabolic disorders (Metabolism and nutrition disorders) | 3 (3) | 3 (3)
Hematologic malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 6 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omidubicel (N=52) | Unmanipulated CBU(s) (N=56)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 5 (8)
Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 17 (18) | 21 (22)
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrointestinal Toxicity (Gastrointestinal disorders) | 40 (42) | 48 (51)
Vomiting (Gastrointestinal disorders) | 33 (33) | 40 (40)
Asthenia (General disorders) | 31 (32) | 42 (44)
Mucosal Inflammation (General disorders) | 39 (40) | 47 (47)
Edema (General disorders) | 24 (24) | 37 (37)
Pain (General disorders) | 41 (42) | 43 (45)
Pyrexia (General disorders) | 42 (42) | 54 (54)
veno-occlusive liver disease (Hepatobiliary disorders) | 2 (2) | 5 (5)
acute graft-versus-host-disease (Immune system disorders) | 18 (18) | 12 (12)
Chronic Graft-versus-host-disease (Immune system disorders) | 0 (0) | 3 (3)
Hypersensitivity (Immune system disorders) | 4 (4) | 10 (10)
Cystitis (Infections and infestations) | 12 (12) | 11 (11)
CMV Infection (Infections and infestations) | 5 (5) | 3 (3)
Herpes infection (Infections and infestations) | 3 (3) | 2 (2)
Human Herpesvirus 6 infection (Infections and infestations) | 5 (5) | 3 (3)
Lower respiratory infection (Infections and infestations) | 5 (5) | 6 (6)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Septic shock (Infections and infestations) | 1 (1) | 8 (9)
Staphylococcal infection (Infections and infestations) | 3 (3) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 5 (5) | 10 (10)
Transplant Failure (Injury, poisoning and procedural complications) | 3 (3) | 5 (5)
Transaminases increased (Investigations) | 4 (4) | 1 (1)
Weight decreased (Investigations) | 23 (23) | 21 (21)
Dehydration (Metabolism and nutrition disorders) | 11 (11) | 10 (10)
Hyperglycemia (Metabolism and nutrition disorders) | 4 (5) | 8 (11)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 3 (4)
Hypokalemia (Metabolism and nutrition disorders) | 6 (6) | 5 (5)
Fluid overload (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 5 (5)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 16 (16) | 22 (22)
Disease recurrence (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 6 (6)
Syncope (Nervous system disorders) | 3 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 15 (15) | 21 (23)
Depression (Psychiatric disorders) | 13 (13) | 16 (16)
Insomnia (Psychiatric disorders) | 24 (24) | 26 (26)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 3 (3)
Cystitis hemorrhagic (Renal and urinary disorders) | 0 (0) | 3 (3)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 26 (27)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 16 (16)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 23 (23)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 5 (5)
Hemorrhage (Vascular disorders) | 14 (14) | 20 (20)
Hypertension (Vascular disorders) | 29 (29) | 37 (37)
Hypotension (Vascular disorders) | 16 (16) | 19 (19)
Arrhythmia (Cardiac disorders) | 24 (24) | 30 (32)
Dry eye (Eye disorders) | 6 (6) | 10 (11)
Vision blurred (Eye disorders) | 3 (3) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 10 (10) | 16 (16)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Constipation (Gastrointestinal disorders) | 12 (12) | 21 (21)
Dyspepsia (Gastrointestinal disorders) | 12 (12) | 12 (12)
Hemorrhoids (Gastrointestinal disorders) | 1 (1) | 3 (3)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2)
Chills (General disorders) | 19 (19) | 32 (32)
Bacteremia (Infections and infestations) | 0 (0) | 2 (2)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 7 (7)
Dizziness (Nervous system disorders) | 10 (10) | 13 (13)
Dysgeusia (Nervous system disorders) | 15 (15) | 9 (9)
Somnolence (Nervous system disorders) | 7 (7) | 12 (12)
Tremor (Nervous system disorders) | 8 (8) | 12 (12)
Cough (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 30 (30)
Dry skin (Skin and subcutaneous tissue disorders) | 21 (21) | 10 (10)
Pruritus (Skin and subcutaneous tissue disorders) | 21 (21) | 28 (28)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 16 (16) | 15 (15)
Skin ulcer (Skin and subcutaneous tissue disorders) | 4 (4) | 6 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review/comment at least 30 days before publication submission. At Sponsor request, site will withhold publication another 60 days to allow for patent application or other measures Sponsor deems appropriate to establish & preserve its proprietary rights. Results publication made as part of those obtained by all sites performing protocol. Site free to publish based on its study results after publication of multi-center results or one year after completion/termination of site study.

DOCUMENTS (2):
  • Study Protocol (2019-01-22): https://cdn.clinicaltrials.gov/large-docs/99/NCT02730299/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT02730299/SAP_001.pdf